CLINICAL TRIAL: NCT02079441
Title: Immune Function in Offsprings of Females With Inflammatory Bowel Disease (IBD) Treated With Anti-TNF Medications During Pregnancy
Brief Title: Immune Function in Offsprings of Females With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Schneider Children's Hospital (Other); Tel Aviv Medical Center (Other); Shaare Zedek Medical Center (Other); Assaf-Harofeh Medical Center (Other Government); Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Batia Weiss, Director, Pediatric Gastroenterology and Nutrition Unit, Sheba Medical Center
Other Study IDs: SHEBA-13-0613-BW-CTIL
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: Anti- TNF; inflammatory bowel disease; pregnancy; infant; immunity; Immune function
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants, IBD, anti TNF, pregnancy: Infants of mothers with anti-TNF in pregnancy
- infants, IBD, pregnancy, medications: Infants of mothers with non anti TNFin pregnancy

SUMMARY:
1. To evaluate the immune response to vaccines in infants of IBD patients treated with anti-TNF medications during pregnancy compared to infants of IBD mother not treated with anti-TNF medications.
2. To evaluate the immune function of B and T cells at 3 months and one year of age in infants of IBD patients treated with anti-TNF medications during pregnancy compared to infants of non anti-TNF treated mothers.

The secondary aims are to follow anti TNF drug levels in infants born to IBD patients treated with anti-TNF medications during pregnancy and to evaluate the risk of infections during the first year of life in this population, compared to children of IBD patients not treated with anti-TNF medications during pregnancy.

Significance -The results of this study have the potential to change clinical practice of anti TNF treatment during pregnancy and the follow-up of infants born to these patients

DETAILED DESCRIPTION:
1. We aim to evaluate the immune response to vaccines in infants of IBD patients treated with anti-TNF medications during pregnancy compared to infants of IBD mother not treated with anti-TNF medications.

2 WE aim to evaluate the immune function of B and T cells at 3 months and one year of age in infants of IBD patients treated with anti-TNF medications during pregnancy compared to infants of non anti-TNF treated mothers.

Our secondary aims are to follow anti TNF drug levels in infants born to IBD patients treated with anti-TNF medications during pregnancy and to evaluate the risk of infections during the first year of life in this population, compared to children of IBD patients not treated with anti-TNF medications during pregnancy.

The results of this study have the potential to change clinical practice of anti TNF treatment during pregnancy and the follow-up of infants born to these patients

ELIGIBILITY:
Inclusion Criteria:

1. Children born to mothers with IBD who were treated with ant-TNF medications, other medications or not medically treated for IBD during pregnancy .
2. Regular vaccination for hepatitis B at birth, 1 and 6 months of age and other scheduled non-live vaccines at 2,4, and 6 months of age.
3. Inform consent signed by the parents.

Exclusion Criteria:

1. Children with intrauterine or perinatal infections, congenital diseases or malformations.
2. Absence of immunization records.
3. Known immune deficiency of mother and/or child. 4. Mothers with hepatitis B

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a multicenter prospective controlled trial. The study population includes infants born to mothers with IBD, divided into two groups: Study group- infants of IBD patients treated with anti-TNF during pregnancy. Control group- infants of IBD patients treated with non-anti TNF medications during pregnancy.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Antibodies to vaccine agents at age 12 months. 2. Immunoglobulin levels, B and T cell production (IgG subclasses, T cell subpopulation numbers) and function (response to mitogens and antigens) at age 3 months and 1 year | 12 months

SECONDARY OUTCOMES:
Anti TNF drug level in cord blood | birth
Infection number and type during the first year of life | 12 months
Antibiotic use in the first year | 12 months
Breast feeding influence (with and without additional medications) on the immune function of the children | 12 months
  Not performed

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No